CLINICAL TRIAL: NCT00032422
Title: Acupuncture in Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT000671-01 (NIH)
Record Dates: First submitted 2002-03-20; First posted 2002-03-22 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Congestive Heart Failure
Keywords: Acupuncture; Heart Failure; Autonomic nervous system
MeSH Terms: conditions — Heart Failure | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to determine if acupuncture decreases adrenaline levels in heart failure, thereby potentially improving survival and quality of life.

DETAILED DESCRIPTION:
Acupuncture is used to lower blood pressure in patients with hypertension, and to relieve angina in patients with coronary artery disease. While the biological mechanisms of acupuncture analgesia have been studied intensely in animals and humans, the biological mechanisms for modulation of the cardiovascular system in humans remain largely unexplored. Acupuncture at traditional acupoints, and at nonacupoints, decreases the blood pressure response during mental stress in normal humans. This depressor effect cannot be fully explained by a decline in muscle sympathetic nerve activity (MSNA). Further, in humans with heart failure (HF) in whom MSNA is elevated, we have preliminary data that acupuncture significantly decreases the MSNA response during mental stress. The following hypotheses will be tested: 1) acupuncture, performed at traditional acupoints and non-acupoints in normal humans, stimulates skeletal muscle afferent neurons causing a release of endogenous opioids, which oppose sympathetic excitation and vasoconstriction in visceral vascular beds, such as the kidney; 2) in humans with HF in whom MSNA is elevated and renal vasoconstriction is the rule, acupuncture utilizes similar mechanisms as in normal humans to produce exaggerated inhibition of MSNA and reflex renal vasoconstriction. Positron emission tomography and microneurography will be utilized to answer the following questions in normal humans and patients with heart failure: 1. Is acupuncture attenuation of BP during mental stress mediated by a decrease in renal vasoconstriction? 2. Is acupuncture sympathoinhibitory? 3. Is acupuncture modulation of the autonomic nervous system mediated by muscle afferents? 4. Is acupuncture modulation of the autonomic nervous system mediated by activation of endogenous opioids? Understanding the mechanisms of acupuncture modulation of the autonomic nervous system in humans may help clarify its role as a therapeutic modality in cardiovascular diseases, such as heart failure.

ELIGIBILITY:
* Chronic congestive heart failure class II-III
* No unstable angina
* No myocardial infarction within 3 months
* No peripheral neuropathy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-07; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Holly R Middlekauff, MD, Principal Investigator — University of California, Los Angeles; KaKit Hui, MD — UCLA East/West Medical Center
Locations (1):
- UCLA School of Medicine, Los Angeles, California, United States

REFERENCES:
- [Background] Middlekauff HR, Yu JL, Hui K. Acupuncture effects on reflex responses to mental stress in humans. Am J Physiol Regul Integr Comp Physiol. 2001 May;280(5):R1462-8. doi: 10.1152/ajpregu.2001.280.5.R1462. PMID 11294769